CLINICAL TRIAL: NCT04545944
Title: An Open-Label, Fixed Sequence, Clinical Drug Interaction Study to Evaluate the Time-Dependent Inhibition Potential of Vonoprazan on a Sensitive CYP3A4 Substrate, Midazolam, in Healthy Volunteers
Brief Title: Evaluation of Effect of Vonoprazan on Midazolam Pharmacokinetics in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phathom Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VONO-101
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Results first posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteers
Keywords: vonoprazan; midazolam
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Midazolam single doses / Vonoprazan multiple doses (Experimental): Single oral doses of 2 mg of midazolam syrup on Day 1 and Day 9 and twice daily (BID) doses of 20 mg vonoprazan oral tablets on Days 2 through 10
  Interventions: Drug: Vonoprazan; Drug: Midazolam

INTERVENTIONS:
Drug: Vonoprazan — 20 mg tablets administered orally
Drug: Midazolam — 2 mg syrup administered orally

SUMMARY:
To determine the time-dependent inhibition potential of repeated doses of oral vonoprazan on the pharmacokinetics (PK) of a single oral dose of midazolam, a sensitive cytochrome P450 3A4 (CYP3A4) substrate, in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Inclusion Criteria:

1. The participant is male or female 18 to 45 years of age, inclusive, at Screening.
2. The participant has a body mass index (BMI) 18 to 30 kg/m2, inclusive, and body weight >50 kg at Screening.
3. The participant is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings at Screening.
4. Female participants of childbearing potential who may be sexually active with a non-sterilized male partner must use an acceptable method of birth control (ie, diaphragm with spermicide, intrauterine device, condom with foam or vaginal spermicide, oral contraceptives, or abstinence) from the signing of informed consent until 4 weeks after the last dose of study drug or be surgically sterile (ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or postmenopausal (defined as amenorrhea for 12 consecutive months and documented plasma follicle-stimulating hormone [FSH] level >40 IU/mL).
5. Female participants must have a negative pregnancy test at Screening and Check-in.
6. The participant agrees to comply with all protocol requirements.
7. The participant is able to provide written informed consent.

Exclusion Criteria:

1. The participant has a history of any clinically significant neurological, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urological, hematological, or endocrine disease or other abnormality that may affect the ability of the subject to participate in the study.
2. The participant has a positive test result for coronavirus disease 2019 (COVID-19), hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus type 1 or 2 antibodies at Screening.
3. The participant has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 × the upper limit of normal (ULN) or total bilirubin >1.5 × ULN (with the exception of Gilbert's syndrome) at Screening or Check-in.
4. The participant has serum creatinine >1.2 mg/dL or blood urea nitrogen >20 mg/dL at Screening or Check-in.
5. The participant has any acute laboratory abnormality at Screening that precludes participation in the study, in the opinion of the investigator.
6. The participant has a current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome and asymptomatic gallstones).
7. The subject has used any prescription (excluding hormonal birth control) or over-the-counter medications (including CYP3A4 inducers) except paracetamol (up to 2 g per day), including herbal or nutritional supplements, within 14 days (or 5 half-lives) before the first dose of study drug or throughout the study.
8. The subject has consumed grapefruit or grapefruit juice, Seville orange or Seville orange-containing products (eg, marmalade), or food products that may be CYP3A4 inhibitors (eg, vegetables from the mustard green family [kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard] and charbroiled meats) within 7 days (or 5 half-lives) before the first dose of study drug or throughout the study.
9. The subject has consumed caffeine or xanthine-containing products within 48 hours (or 5 half-lives) before the first dose of study drug or throughout the study.
10. The subject is a smoker or has used nicotine or nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) within 6 months before the first dose of study drug.
11. The subject has a history of alcohol abuse or drug addiction within the last year, excessive alcohol consumption (regular alcohol intake >21 units per week for male subjects and >14 units of alcohol per week for female subjects; 1 unit is equal to approximately 1/2 pint [200 mL] of beer, 1 small glass [100 mL] of wine, or 1 measure.
12. The subject has a positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking) at Screening or Check-in.
13. The subject is involved in strenuous activity or contact sports within 24 hours before the first dose of study drug or throughout the study.
14. The subject has donated blood or blood products >450 mL within 30 days before the first dose of study drug.
15. The subject has a history of relevant drug and/or food allergies (ie, allergy to midazolam, vonoprazan, or their excipients [including cherries] or any significant food allergy that could preclude a standard diet in the clinical unit).
16. The subject has received study drug in another investigational study within 30 days of dosing.
17. Female subject is pregnant or lactating, intends to become pregnant before, during, or within 4 weeks after participating in this study, or intends to donate ova during this time period.
18. The subject has a history of acute narrow-angle glaucoma.
19. In the opinion of the investigator, the subject is not suitable for entry into the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Phathom Pharmaceuticals, Inc.
Locations (1):
- PPD Development, LP, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 participants were enrolled at a single study center in the United States.
Pre-assignment Details: 32 participants were screened, 12 of which were screen failures. The remaining 20 were enrolled and received study treatment.
Groups:
- All Participants: All participants were administered single oral doses of 2 milligrams (mg) of midazolam syrup on Day 1 and Day 9 and twice per day (BID) oral doses of 20 mg vonoprazan tablets on Days 2 through 10.
Period: Overall Study
Arm/Group | All Participants
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants were administered single oral doses of 2 mg of midazolam syrup on Day 1 and Day 9 and BID oral doses of 20 mg vonoprazan tablets on Days 2 through 10.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (7.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 7
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Last Quantifiable Concentration (AUC0-t) of Midazolam
Description: AUC0-t was measured for midazolam alone on Day 1 and for midazolam administered with vonoprazan on Day 9.
Time Frame: Day 1 (midazolam alone): Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post-dose; Day 9 (midazolam and vonoprazan): Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post-dose
Population: The pharmacokinetics (PK) population included participants who received at least one dose of study drug and had sufficient concentration data to support accurate estimation of at least one PK parameter. Participants who experienced vomiting within two times the median time to maximum observed plasma concentration (Tmax) after midazolam dosing were excluded from the PK analysis.
Measure: Mean (Standard Deviation); unit: Nanogram Hours per Milliliter (ng•h/mL)
Groups:
- Midazolam Alone: Participants were administered a single oral dose of 2 mg of midazolam syrup on Day 1.
- Midazolam With Vonoprazan: Participants were administered a single oral dose of 2 mg of midazolam syrup on Day 9 and BID oral doses of 20 mg vonoprazan tablets on Day 2 to Day 10.
Arm/Group | Midazolam Alone | Midazolam With Vonoprazan
Number analyzed (Participants) | 20 | 20
Nanogram Hours per Milliliter (ng•h/mL) | 24.2 (8.76) | 50.7 (39.8)
Statistical Analysis 1: Comparison: Midazolam Alone vs Midazolam With Vonoprazan; A linear mixed model with treatment as a fixed effect and participant as a random effect was performed on the natural log-transformed values to assess the effect of vonoprazan on the PK of midazolam; Test type: Other; Geometric Least Squares Mean Ratio = 192.4, 90% CI 2-sided [152.8 to 242.4]

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Midazolam
Description: AUC0-inf was measured for midazolam alone on Day 1 and for midazolam administered with vonoprazan on Day 9.
Time Frame: as for outcome 1
Population: The PK population included participants who received at least one dose of study drug and had sufficient concentration data to support accurate estimation of at least one PK parameter. Participants who experienced vomiting within two times the median time to maximum observed plasma concentration (Tmax) after midazolam dosing were excluded from the PK analysis.
Measure: Mean (Standard Deviation); unit: Nanogram Hours per Milliliter (ng•h/mL)
Arm/Group | Midazolam Alone | Midazolam With Vonoprazan
Number analyzed (Participants) | 20 | 20
Nanogram Hours per Milliliter (ng•h/mL) | 25.5 (9.00) | 52.3 (39.8)
Statistical Analysis 1: Comparison: Midazolam Alone vs Midazolam With Vonoprazan; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric Least Squares Mean Ratio = 188.9, 90% CI 2-sided [150.6 to 236.9]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Midazolam
Description: Cmax was measured for midazolam alone on Day 1 and for midazolam administered with vonoprazan on Day 9.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Nanograms per Milliliter (ng/mL)
Arm/Group | Midazolam Alone | Midazolam With Vonoprazan
Number analyzed (Participants) | 20 | 20
Nanograms per Milliliter (ng/mL) | 10.3 (3.61) | 20.3 (9.55)
Statistical Analysis 1: Comparison: Midazolam Alone vs Midazolam With Vonoprazan; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric Least Squares Mean Ratio = 193.4, 90% CI 2-sided [160.5 to 233.1]

ADVERSE EVENTS:
Time Frame: Day 1 to Day 25
Description: The safety population included all participants who received at least one dose of study drug. Treatment-emergent adverse events were summarized by treatment (midazolam alone, vonoprazan alone and midazolam with vonoprazan) and an event was assigned to the last treatment the participant received when the event occurred.
Groups:
- Vonoprazan Alone: Participants were administered BID oral doses of 20 mg vonoprazan tablets alone on Day 2 through Day 8.
- Midazolam With Vonoprazan: Participants were administered single oral doses of 2 mg of midazolam syrup on Day 9 and BID oral doses of 20 mg vonoprazan tablets on Days 9 and 10.
Arm/Group | Midazolam Alone | Vonoprazan Alone | Midazolam With Vonoprazan
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 4/20 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam Alone (N=20) | Vonoprazan Alone (N=20) | Midazolam With Vonoprazan (N=20)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling drunk (General disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PPD cannot publish data from a Phathom trial (or assist a third party with a publication) that includes any vonoprazan data without consent.

DOCUMENTS (2):
  • Study Protocol (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/44/NCT04545944/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT04545944/SAP_001.pdf